CLINICAL TRIAL: NCT06735222
Title: Hydroxytyrosol Bioavailability in Humans: A Comparative Study of Three EPA-Enriched Formulations
Brief Title: Bioavailability of Hydroxytyrosol in Humans Co-administered With EPA
Acronym: HydroxyOmegaBd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Olivenova Health Sl (Unknown)
Responsible Party: Principal Investigator, María Raquel Mateos Briz, Investigator, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HYDROXYOMEGA-BIOAVAILABILITY
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Young
Keywords: Bioavailability; hydroxytyrosol; nutraceutical; omega-3; nutrikinetics
MeSH Terms: interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Intervention Model Description: Acute, randomized, cross-over, controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HT-Ac → HT-EPA → Oleacore® (Experimental): Group 1 will consume HT-Ac in the first week, HT-EPA in the second week and Oleacore® in the third week.
  Interventions: Dietary Supplement: Hydroxytyrosol acetate (HT-Ac); Dietary Supplement: Hydroxytyrosol eicosapentanoate (HT-EPA); Dietary Supplement: Oleacore®
- HT-EPA → Oleacore® → HT-Ac (Experimental): Group 2 will consume HT-EPA in the first week, Oleacore® in the second week and HT-Ac in the third week.
  Interventions: Dietary Supplement: Hydroxytyrosol acetate (HT-Ac); Dietary Supplement: Hydroxytyrosol eicosapentanoate (HT-EPA); Dietary Supplement: Oleacore®
- Oleacore® → HT-Ac → HT-EPA (Experimental): Group 3 will consume Oleacore® in the first week, HT-Ac in the second week and HT-EPA in the third week.
  Interventions: Dietary Supplement: Hydroxytyrosol acetate (HT-Ac); Dietary Supplement: Hydroxytyrosol eicosapentanoate (HT-EPA); Dietary Supplement: Oleacore®

INTERVENTIONS:
Dietary Supplement: Hydroxytyrosol acetate (HT-Ac) — Hydroxytyrosol acetate (15 mg) orally co-administered with 2 g EPA
Dietary Supplement: Hydroxytyrosol eicosapentanoate (HT-EPA) — Oral intake of hydroxytyrosol eicosapentanoate (15 mg) solubilized in an EPA-enriched oil matrix.
Dietary Supplement: Oleacore® — Oleacore® (containing 15 mg of hydroxytyrosol) orally co-administered with 2 g EPA

SUMMARY:
The primary objective of this study is to evaluate the optimal formulation of a natural nutraceutical whose daily consumption at nutritional doses may confer benefits for cardiovascular health. This nutraceutical combines an omega-3 fatty acid (eicosapentaenoic acid, EPA) with hydroxytyrosol (a potent antioxidant found in olives and extra virgin olive oil). The study will allow to compare how and to what extent hydroxytyrosol is absorbed when co-administered the omega-3 fatty acid in capsules across three different formulations.

DETAILED DESCRIPTION:
12 healthy male and female participants will consume various formulations corresponding to three nutraceuticals developed: hydroxytyrosol acetate (HT-Ac), hydroxytyrosol eicosapentanoate (HT-EPA), and hydroxytyrosol extract (Oleacore®) with EPA. One week prior to the intervention, participants will be instructed to refrain from consuming extra virgin olive oil or olives as the primary dietary sources of hydroxytyrosol (wash-out phase). Since three types of nutraceuticals will be evaluated, the study will take place over three separate days, with one week between each intervention.

On each intervention day, following an overnight fast, volunteers will randomly consume one of the nutraceuticals. A polyphenol-free diet will be provided during the 24 hours after the nutraceutical intake.

Blood samples will be collected right before the nutracetical intake at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-consumption. Urine samples will also be collected in 24-hour collection containers containing 0.5 g of ascorbic acid, at the following intervals: -2 to 0 hours (baseline), 0-3 hours, 3-6 hours, 6-10 hours, and 10-24 hours. All of these samples will be stored at -80ºC until analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 45 years old
* Body Mass Index (BMI): 18 to 25 kg/m²

Exclusion Criteria:

* Presence of chronic illnesses
* Currently undergoing pharmacological treatment
* Smoking
* Pregnancy
* Following a vegetarian or vegan diet

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Targeted and untargeted metabolomics | Up to 6 months
  The determination of HT metabolites in plasma and urine of the healthy volunteers following the consumption of nutraceuticals will be carried out using both targeted and untargeted metabolomics through high-performance liquid chromatography coupled to an Accurate-Mass Quadrupole Time-of-Flight (QToF) with ESI-Jet Stream Technology (HPLC-ESI-QToF, Agilent Technologies). Additionally, three types of nutraceuticals (EPA-HT, EPA+HT-Ac and EPA-Oleacore®) will be tested in order to evaluate the HT bioavailability comparatively.

SECONDARY OUTCOMES:
ox-LDL as marker of oxidative status | Up to 2 months
  Differences between non-supplemented subjects and those supplemented with HT-Ac, HT-EPA, and Oleacore®, analyzed across different blood collection times.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Mateos Briz Tenured Scientist, Principal Investigator — 1
Locations (1):
- Ictan-Csic, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No